CLINICAL TRIAL: NCT01190839
Title: Prospective, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial Comparing REMICADE (Infliximab) and Placebo in the Prevention of Recurrence in Crohn's Disease Patients Undergoing Surgical Resection Who Are at Increased Risk of Recurrence
Brief Title: A Multicenter Trial Comparing REMICADE (Infliximab) and Placebo in the Prevention of Recurrence in Crohn's Disease (CD) Patients Undergoing Surgical Resection Who Are at an Increased Risk of Recurrence
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study is terminated as per Sponsor's Decision.
Sponsor: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR017080; REMICADECRD3001 (Other: Janssen Biotech Inc.); 2010-018431-18 (EudraCT Number); PREVENT (Other: Janssen Biotech Inc.)
Record Dates: First submitted 2010-08-12; First posted 2010-08-30 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2015-12

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Inflammatory Bowel Disease; infliximab; TNF-alpha
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infliximab (Experimental): Infliximab Type=equal unit=mg number=5 form=intravenous infusion route=intravenous use once every 8 weeks
  Interventions: Biological: Infliximab
- Placebo (Placebo Comparator): Placebo Type=equal unit=mg number=5 form=intravenous infusion route=intravenous use once every 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Infliximab — Type=equal, unit=mg, number=5, form=intravenous infusion, route=intravenous use, once every 8 weeks
  Arms: Infliximab
Drug: Placebo — Type=equal, unit=mg, number=5, form=intravenous infusion, route=intravenous use, once every 8 weeks
  Arms: Placebo

SUMMARY:
REMICADE (infliximab) is a drug used to treat active Crohn's disease and is being tested in an experiment to see if it may be useful in preventing relapse of Crohn's disease after surgical resection. This study will compare the effects (both good and bad) of REMICADE (infliximab) to those of placebo. Placebo looks like the drug being studied but has no active ingredients.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effects of REMICADE (infliximab) in preventing relapse of Crohn's disease after surgical resection. Patients will be assigned to a group that will initially receive either infliximab or placebo. Each patient who is allowed to join the study is put into a group by chance (randomly), like flipping a coin. There is a possibility that patients can receive both the study drug and placebo at different times in the study. If a patient is initially randomized to receive placebo, and their study doctor confirms that they have had a return of active Crohn's Disease symptoms, they can receive infliximab. If a patient is initially randomized to receive infliximab, and their study doctor confirms that they are experiencing symptoms of Crohn's Disease, they may receive an increase in their infliximab dose. Infusions will be administered at Week 0 and then every 8 weeks thereafter through Week 200. The study will use a measure of Crohn's Disease activity that will be evaluated at each visit and at any time the patient has symptoms suggestive of their disease getting worse in order to capture recurrence. During the study, patients who meet the study definition of clinical recurrence will be eligible to have a blinded infliximab dose increase of 5 mg/kg. In other words, patients receiving placebo would receive infliximab 5 mg/kg, and patients receiving infliximab 5 mg/kg would have a dose increase to 10 mg/kg. Approximately 175 sites will be utilized, and approximately 290 patients will be enrolled. The interval between the first and last dose of study agent is 200 weeks. The planned duration of study participation is a maximum of 209 weeks (with a 1-week screening period, a 200-week treatment period, and a final study visit at Week 208). Group I (infliximab infusions): infliximab (5 mg/kg) will be administered by intravenous (IV) infusion at Week 0 and every 8 weeks thereafter through Week 200. Group II (placebo infusions): placebo will be administered by IV infusion at Week 0 and every 8 weeks thereafter through Week 200

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of CD confirmed by endoscopic, histologic and/or radiologic studies prior to resection or by tissue obtained at resection
* Have undergone an ileocolonic surgical resection
* Patients must also be at an increased risk of recurrence of active CD
* Patients must not have previously discontinued infliximab as a result of tolerability issues or they must be naive to treatment with infliximab. Provided patients meet the above criteria pertaining to infliximab, they are eligible to enroll if they received prior treatment with adalimumab and/or certolizumab
* Patients must undergo screening for HBV
* Baseline CDAI < 200
* Have adequate blood and liver test values

Exclusion Criteria:

* Have a history of latent or active granulomatous infection, including histoplasmosis or coccidioidomycosis, prior to screening
* Have a chest radiograph within 3 months prior to the first infusion of study agent that shows a clinically significant abnormality, such as a malignancy or infection, or any abnormalities suggestive of TB
* Have macroscopically active CD which was not resected at the time of surgery
* Do not meet the criteria for being at an increased risk of postoperative recurrence of active CD as outlined in the inclusion criteria
* Have evidence of an active infection at the time of randomization or have had a serious infection not related to CD (e.g., hepatitis, pneumonia, or pyelonephritis), within 6 months prior to screening
* Have or have had an opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening
* Have any known malignancy or history of malignancy within the 5-year period prior to screening (with the exception of squamous or basal cell carcinoma of the skin that has been completely excised without evidence of recurrence)
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2010-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Biotech Inc. Clinical Trial, Study Director — Janssen Biotech, Inc.
Locations (142):
- United States (62):
  - Birmingham, Alabama
  - La Jolla, California
  - Orange, California
  - Redwood City, California
  - San Diego, California
  - Littleton, Colorado
  - Glastonbury, Connecticut
  - Middletown, Connecticut
  - New Haven, Connecticut
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Naples, Florida
  - Weston, Florida
  - Winter Park, Florida
  - Decatur, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Clive, Iowa
  - Iowa City, Iowa
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Chevy Chase, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Troy, Michigan
  - Plymouth, Minnesota
  - Rochester, Minnesota
  - Lees Summit, Missouri
  - Lebanon, New Hampshire
  - Morristown, New Jersey
  - Great Neck, New York
  - New York, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Grapevine, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Charlottesville, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Tacoma, Washington
  - Madison, Wisconsin
- Australia (6):
  - Adelaide
  - Brisbane
  - Fremantle
  - Herston
  - Malvern
  - Nambour
- Austria (3):
  - Graz
  - Salzburg
  - Vienna
- Belgium (6):
  - Bonheiden
  - Brussels
  - Ghent
  - Leuven
  - Liège
  - Roeselare
- Canada (12):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Brandon, Manitoba
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Guelph, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Lévis, Quebec
  - Montreal, Quebec
  - Québec, Quebec
- Czechia (2):
  - Litoměřice
  - Prague
- France (11):
  - Bordeaux
  - Caen
  - Grenoble
  - Lille
  - Marseille
  - Nantes
  - Nice
  - Paris
  - Pessac
  - Rouen
  - Vandœuvre-lès-Nancy
- Germany (12):
  - Berlin
  - Erlangen
  - Hamburg
  - Hanover
  - Heidelberg
  - Herne
  - Kiel
  - Lÿneburg
  - Mannheim
  - München
  - Münster
  - Tübingen
- Hungary (4):
  - Békéscsaba
  - Budapest
  - Debrecen
  - Pécs
- Israel (3):
  - Jerusalem
  - Petah Tikva
  - Tel Aviv
- Netherlands (6):
  - Almere Stad
  - Amsterdam
  - Amsterdam-Zuidoost
  - Leiden
  - Maastricht
  - Rotterdam
- New Zealand (5):
  - Auckland
  - Christchurch
  - Dunedin
  - Hamilton
  - Wellington
- Poland (3):
  - Lodz
  - Warsaw
  - Wroclaw
- United Kingdom (7):
  - Cambridge
  - Cardiff
  - London
  - Manchester
  - Norwich
  - Nottinghamshirecc
  - Oxford

REFERENCES:
- [Derived] Regueiro M, Feagan BG, Zou B, Johanns J, Blank MA, Chevrier M, Plevy S, Popp J, Cornillie FJ, Lukas M, Danese S, Gionchetti P, Hanauer SB, Reinisch W, Sandborn WJ, Sorrentino D, Rutgeerts P; PREVENT Study Group. Infliximab Reduces Endoscopic, but Not Clinical, Recurrence of Crohn's Disease After Ileocolonic Resection. Gastroenterology. 2016 Jun;150(7):1568-1578. doi: 10.1053/j.gastro.2016.02.072. Epub 2016 Mar 3. PMID 26946343

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants randomized to receive placebo at Week 0 and then every 8 weeks thereafter through Week 200.
- Infliximab 5 mg/kg: Participants randomized to receive Infliximab 5 milligram per kilogram (mg/kg) at Week 0 and then every 8 weeks thereafter through Week 200.
Period: Overall Study
Arm/Group | Placebo | Infliximab 5 mg/kg
Started | 150 | 147
Treated | 148 | 143
Completed | 0 | 0
Not Completed | 150 | 147
Not completed — Adverse Event | 32 | 41
Not completed — Protocol Violation | 2 | 2
Not completed — Lost to Follow-up | 7 | 1
Not completed — Death | 1 | 0
Not completed — Trial stopped by Sponsor | 71 | 68
Not completed — Undefined | 35 | 31
Not completed — Randomized but not treated | 2 | 4

BASELINE CHARACTERISTICS:
Population: Analysis population included all the participants who were randomly assigned to receive 1 of the study treatments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Infliximab 5 mg/kg | Total
Number analyzed (Participants) | 150 | 147 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (12.41) | 37.1 (13.49) | 36.3 (12.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 70 | 139
  Male | 81 | 77 | 158

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Recurrence (CR) of Crohn's Disease (CD) Prior to or at Week 76
Description: CR criteria:1) A >=70-point increase from baseline in CDAI score [in general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities];2)A CDAI score >=200;3)Evidence of endoscopic recurrence [ileal Rutgeerts score of >=i2 at anastomotic site or its equivalent elsewhere in GI tract] and 4)A negative stool test for C. difficile toxin (if, in the opinion of the investigator, the participant's symptoms are predominantly diarrheal); or at least 1 of followings:1) developing a new draining external fistula;2)re-opening and draining of a previously existing external fistula;3)developing a new internal fistula;4)developing a new perianal abscess or 5)developing a new intra-abdominal abscess more than 3 months after date of index surgery. In addition, participants who had a treatment failure [initiated a prohibited CD medication, had prohibited use of CD medication, or had surgery for CD] before or at Week 76 were considered to have clinical recurrence.
Time Frame: Baseline up to Week 76
Population: Analysis population included all the participants who were randomly assigned to receive 1 of the study treatments.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Infliximab 5 mg/kg
Number analyzed (Participants) | 150 | 147
percentage of participants | 20.0 | 12.9
Statistical Analysis 1: Comparison: Placebo vs Infliximab 5 mg/kg; Test type: Superiority or Other; p = 0.097, Cochran-Mantel-Haenszel chi-square test — p-value was based on the Cochran-Mantel-Haenszel chi-square test stratified by the number of risk factors for recurrence of active CD and baseline use of an immunomodulator

2. Secondary Outcome: Percentage of Participants With Endoscopic Recurrence of CD Prior to or at Week 76
Description: Endoscopic recurrence is defined as an ileal Rutgeert's score of >= i2 either at the anastomotic site or elsewhere in the gastrointestinal tract. In addition, participants who had a treatment failure (initiated a prohibited CD medication, had a prohibited use of a CD medication, or had a surgery for CD) prior to Week 76, and who developed a new draining external fistula or re-opening and draining of a previously existing external fistula or developed a new internal fistula, new perianal abscess or new intra-abdominal abscess more than 3 months after the date of the index surgery were considered to have had endoscopic recurrence prior to or at Week 76.
Time Frame: Baseline up to Week 76
Population: Analysis population included all the participants who were randomly assigned one of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Infliximab 5 mg/kg
Number analyzed (Participants) | 150 | 147
percentage of participants | 60.0 | 30.6
Statistical Analysis 1: Comparison: Placebo vs Infliximab 5 mg/kg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With Clinical Recurrence (CR) of Crohn's Disease (CD) Prior to or at Week 104
Description: CR criteria:1) A >=70-point increase from baseline in CDAI score [in general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities];2)A CDAI score >=200;3)Evidence of endoscopic recurrence [ileal Rutgeerts score of >=i2 at anastomotic site or its equivalent elsewhere in GI tract] and 4)A negative stool test for C. difficile toxin (if, in the opinion of the investigator, the participant's symptoms are predominantly diarrheal); or at least 1 of followings:1) developing a new draining external fistula;2)re-opening and draining of a previously existing external fistula;3)developing a new internal fistula;4)developing a new perianal abscess or 5)developing a new intra-abdominal abscess more than 3 months after date of index surgery. In addition, participants who had a treatment failure [initiated a prohibited CD medication, had prohibited use of CD medication, or had surgery for CD]before or at Week 104 were considered to have clinical recurrence.
Time Frame: Baseline up to Week 104
Population: Analysis population included all the participants who were randomly assigned to receive 1 of the study treatments.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Infliximab 5 mg/kg
Number analyzed (Participants) | 150 | 147
percentage of participants | 25.3 | 17.7
Statistical Analysis 1: Comparison: Placebo vs Infliximab 5 mg/kg; Test type: Superiority or Other; p = 0.098, Cochran-Mantel-Haenszel chi-square test — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline through the final visit (Average weeks of follow-up for placebo, infliximab 5 mg/kg, first placebo then infliximab 5 mg/kg, and first infliximab 5 mg/kg then infliximab 10 mg/kg groups are 114.4, 117.9, 84.0, and 84,3, respectively)
Description: All participants who received at least 1 infusion of study drug. Placebo, Infliximab 5mg/kg includes data up to dose increase. First Placebo Then Infliximab 5 mg/kg, First Infliximab 5 mg/kg Then Infliximab 10 mg/kg includes data from time of dose increase through the final visit.
Groups:
- Placebo: Participants treated with placebo through the final visit or through a protocol defined dose increase. If a participant had a protocol defined dose increase, only safety results prior to the dose increase will be included in this group.
- Infliximab 5 mg/kg: Participants treated with Infliximab 5 mg/kg at any time through the final visit or through a protocol defined dose increase. If a participants had a protocol defined dose increase, only safety results prior to the dose increase will be included in this group.
- First Placebo Then Infliximab 5 mg/kg: Participants had a protocol defined dose increase from Placebo to infliximab 5 mg/kg. Only safety results after start of infliximab were included in this group.
- First Infliximab 5 mg/kg Then Infliximab 10 mg/kg: Participants had a protocol defined dose increase from infliximab 5 mg/kg to infliximab 10 mg/kg. Only safety results after the dose increase were included in this group.
Arm/Group | Placebo | Infliximab 5 mg/kg | First Placebo Then Infliximab 5 mg/kg | First Infliximab 5 mg/kg Then Infliximab 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 36/146 | 32/145 | 5/27 | 2/9
Other Adverse Events (participants affected / at risk) | 122/146 | 121/145 | 18/27 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=146) | Infliximab 5 mg/kg (N=145) | First Placebo Then Infliximab 5 mg/kg (N=27) | First Infliximab 5 mg/kg Then Infliximab 10 mg/kg (N=9)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal Adhesions (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 4 | 1 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal Fistula (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Crohn's Disease (Gastrointestinal disorders) | 5 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileal Stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 3 | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Adverse Drug Reaction (General disorders) | 0 | 1 | 0/21 | 0/6
Malaise (General disorders) | 1 | 0 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Biliary Colic (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0/21 | 0/6
Anaphylactic Reaction (Immune system disorders) | 0 | 1 | 0 | 0
Serum Sickness (Immune system disorders) | 0 | 1 | 0 | 0
Abdominal Abscess (Infections and infestations) | 2 | 0 | 0 | 0
Abdominal Wall Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Anal Abscess (Infections and infestations) | 1 | 0 | 1 | 0
Cytomegalovirus Infection (Infections and infestations) | 2 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Pilonidal Cyst (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia Legionella (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 1 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1
Anastomotic Leak (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Scar (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0/21 | 0/6
Tetany (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lupus-Like Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Radiculitis (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Foetal Death (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Calculus Ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 2 | 0 | 0
Colpocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Maxillofacial Operation (Surgical and medical procedures) | 1 | 0 | 0/21 | 0/6
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 0 | 0
Stoma Site Infection (Infections and infestations) | 0 | 1 | 0 | 0
Anastomotic Stenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post Procedural Diarrhoea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Intestinal Resection (Surgical and medical procedures) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=146) | Infliximab 5 mg/kg (N=145) | First Placebo Then Infliximab 5 mg/kg (N=27) | First Infliximab 5 mg/kg Then Infliximab 10 mg/kg (N=9)
Anaemia (Blood and lymphatic system disorders) | 10 | 8 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 36 | 25 | 4 | 2
Abdominal Symptom (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Crohn's Disease (Gastrointestinal disorders) | 13 | 10 | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 27 | 24 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 10 | 1 | 0
Flatulence (Gastrointestinal disorders) | 7 | 3 | 0/21 | 1/6
Mouth Ulceration (Gastrointestinal disorders) | 1 | 4 | 0 | 2
Nausea (Gastrointestinal disorders) | 16 | 25 | 0 | 2
Toothache (Gastrointestinal disorders) | 5 | 5 | 1 | 1
Vomiting (Gastrointestinal disorders) | 11 | 14 | 0 | 2
Asthenia (General disorders) | 8 | 5 | 1 | 1
Pyrexia (General disorders) | 17 | 22 | 1 | 3
Anal Abscess (Infections and infestations) | 4 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 10 | 7 | 1 | 0
Influenza (Infections and infestations) | 15 | 12 | 0 | 0
Nasopharyngitis (Infections and infestations) | 37 | 37 | 3 | 1
Purulent Discharge (Infections and infestations) | 0 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 21 | 21 | 5 | 3
Urinary Tract Infection (Infections and infestations) | 7 | 4 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 3 | 7 | 2 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Pulmonary Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Body Temperature Increased (Investigations) | 0 | 1 | 2 | 0
Endoscopy Abnormal (Investigations) | 0 | 0 | 0/21 | 1/6
Faecal Calprotectin (Investigations) | 0 | 3 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 | 26 | 4 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 16 | 1 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 1
Dysplastic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dizziness Postural (Nervous system disorders) | 2 | 2 | 0 | 1
Headache (Nervous system disorders) | 31 | 29 | 1 | 0
Lethargy (Nervous system disorders) | 2 | 2 | 0 | 2
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 2 | 0 | 1
Depression (Psychiatric disorders) | 4 | 9 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 7 | 1 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 14 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 10 | 14 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 10 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 9 | 8 | 0 | 2
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 1
Abdominal Distension (Gastrointestinal disorders) | 8 | 8 | 1 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 8 | 8 | 0 | 1
Anal Fistula (Gastrointestinal disorders) | 2 | 1 | 2 | 1
Aphthous Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 7 | 2 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 5 | 5 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 7 | 1 | 1 | 1
Ileal Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 6 | 1 | 1
Adverse Drug Reaction (General disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 10 | 8 | 1 | 0
Infusion Site Extravasation (General disorders) | 1 | 1 | 0 | 1
Local Swelling (General disorders) | 1 | 2 | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 1 | 2 | 0
Conjunctivitis (Infections and infestations) | 2 | 3 | 0 | 1
Gastroenteritis (Infections and infestations) | 8 | 5 | 0 | 0
Gastroenteritis Salmonella (Infections and infestations) | 0 | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 2 | 5 | 1 | 1
Infected Dermal Cyst (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 7 | 9 | 0 | 1
Tooth Abscess (Infections and infestations) | 2 | 2 | 0 | 1
Post Procedural Diarrhoea (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1
Blood Calcium Decreased (Investigations) | 0 | 0 | 0 | 1
Blood Iron Decreased (Investigations) | 1 | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 8 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 3 | 1 | 1
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 3 | 6 | 0 | 1
Restless Legs Syndrome (Nervous system disorders) | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 2 | 2 | 0 | 1
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Pregnancy of Partner (Social circumstances) | 2 | 2 | 2 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 3 | 8 | 1 | 0
Poor Venous Access (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.